CLINICAL TRIAL: NCT01093612
Title: 64 Cu-DOTA-Trastuzumab Positron Emission Tomography in Women With Advanced HER2 Positive Invasive Breast Cancer
Brief Title: Positron Emission Tomography in Women With Advanced HER2-Positive Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09101; NCI-2010-00322 (Registry Identifier: NCI CTRP); BC095002 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2010-03-23; First posted 2010-03-26 (Estimated); Results first posted 2023-03-28 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Stage IV Breast Cancer
Keywords: HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; 64Cu-DOTA-trastuzumab; Biopsy; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): PART ONE: Patients are randomized to 1 of 3 dose levels. Patients undergo a PET scan 24-48 hours after injection of copper Cu 64-DOTA-trastuzumab. PART TWO: Patients undergo a PET scan 24-48 hours after injection of copper Cu 64-DOTA-trastuzumab.
  Interventions: Procedure: positron emission tomography; Radiation: copper Cu 64-DOTA-trastuzumab; Procedure: Biopsy; Other: Immunohistochemistry staining method; Other: laboratory biomarker analysis; Genetic: mutation analysis

INTERVENTIONS:
Procedure: positron emission tomography — PET images performed on a GE Discovery 16 Ste PET-CT scanner
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Radiation: copper Cu 64-DOTA-trastuzumab — 15 mCi of Cu 64-DOTA-trastuzumab, total trastuzumab dose less than 5 mg.
  Other Names: 64Cu-DOTA-trastuzumab
Procedure: Biopsy — Correlative Studies
  Other Names: biopsies
Other: Immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Other: laboratory biomarker analysis — Correlative studies
Genetic: mutation analysis — Correlative studies

SUMMARY:
RATIONALE: Diagnostic procedures, such as copper Cu 64-DOTA-trastuzumab-labeled PET, may help doctors to plan a better treatment

PURPOSE: This pilot trial is studying copper Cu 64-tetra-azacyclododecanetetra-acetic acid (DOTA)-trastuzumab-labeled positron emission tomography (PET) in women with human epidermal growth factor receptor 2 (HER2)-positive breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the dose of pre-administered cold antibody that optimizes image quality of 64Cu-DOTA-trastuzumab PET without increasing the radiation dose to the heart in women with metastatic HER2 positive breast cancer.

II. Determine whether tumor uptake on 64Cu-DOTA-trastuzumab PET correlates with tumor expression of HER2 in women with metastatic disease.

III. Perform an exploratory analysis of the relationship between uptake on 64Cu-DOTA-trastuzumab PET, HER2 overexpression, and inactivation of the PI3K/Akt pathway.

OUTLINE:

This is a part one dose-determining study followed by a part two study. PART ONE: Patients are randomized to 1 of 3 dose levels. Patients undergo a PET scan 24-48 hours after injection of 64 Cu-DOTA-trastuzumab. PART TWO: Patients undergo a PET scan 24-48 hours after injection of 64 Cu-DOTA-trastuzumab at the optimal dose as determined in part one of the study.

ELIGIBILITY:
Eligibility Part I (Determination of the cold dose)

* Participants must be women who have histological confirmation of metastatic invasive breast cancer that has metastasized outside the region of the primary tumor and axilla. Biopsy must be obtained within 28 days prior to study. Patients must have metastatic disease in lung, liver, soft-tissue or bone to qualify for the study (more than one site is permissible).
* At least 1 non-hepatic site of metastasis greater than or equal to 2 cm in mean diameter must be identified in addition to the site that was biopsied.
* The cancer must over express HER2 as determined by IHC and FISH.
* Patients may have received trastuzumab in the adjuvant, neoadjuvant, or metastatic setting, but cannot have received the drug within the prior 2 months.
* Participants must have normal cardiac ejection fraction.

Eligibility Part 2 (correlation of HER2 expression with PET uptake)

* Participants must be women who have histological confirmation of metastatic invasive breast cancer that has metastasized outside the region of the primary tumor and axilla. Biopsy must be obtained within 28 days prior to study. Patients must have metastatic disease in lung, liver, soft-tissue or bone to qualify for the study (more than one site is permissible).
* At least 1 non-hepatic site of metastasis site greater than or equal to 2 cm in mean diameter must be identified in addition to the site that was biopsied.
* Participants with HER2 1+, 2+ and 3+ by IHC are eligible.
* Patients may have received trastuzumab in the adjuvant, neoadjuvant, or metastatic setting, but cannot have received the drug within the prior 2 months.
* Participants must have normal cardiac ejection fraction.

Ineligibility

* Participants who have received trastuzumab within the prior 2 months
* Participants who are not considered candidates for trastuzumab
* Metastatic disease in a single site
* No metastatic site greater than or equal to 2 cm
* Concurrent malignancy other than skin cancer
* Inability to provide informed consent
* Participants who are pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-03-16 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2026-09-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Mortimer, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- HER2+ Patients: HER2+ patients underwent 64Cu-DOTA-trastuzumab injection, preceded by trastuzumab infusion (45 mg). PET/CT was performed 21-25 (day 1) and 47-49 (day 2) hours after 64Cu-DOTA-trastuzumab injection. Radio-label uptake in prominent lesions was measured as SUVmax.
- HER2- Patients: HER2- patients underwent 64Cu-DOTA-trastuzumab injection, preceded by trastuzumab infusion (45 mg). PET/CT was performed 21-25 (day 1) and 47-49 (day 2) hours after 64Cu-DOTA-trastuzumab injection. Radio-label uptake in prominent lesions was measured as SUVmax.
Period: Overall Study
Arm/Group | HER2+ Patients | HER2- Patients
Started | 11 | 7
Completed | 11 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HER2+ Patients | HER2- Patients | Total
Number analyzed (Participants) | 11 | 7 | 18
Age, Continuous [Median (Full Range); unit: years] | 59 [35 to 75] | 61 [40 to 71] | 60 [35 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 2 | 3
  African American | 2 | 0 | 2
  Hispanic | 3 | 3 | 6
  Native American | 1 | 0 | 1
  White Non-Hispanic | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 11 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Tumor Uptake of 64Cu-DOTA-trastuzumab After 24 Hours
Description: Comparison of uptake between the HER2+ and HER2- groups, treating SUVmax measurements for individual tumors as independent observations. Statistical significance of differences in SUVmax between patient groups was assessed via a nonparametric (Wilcoxon rank-sum) test.
  Radiolabel uptake for tumors was measured in terms of single-voxel maximum SUV (SUVmax; SUV = tissue activity per mL x body weight [g]/injected activity decay-corrected to time of scan).
Time Frame: 24 hours after injection of 64 CU-DOTA-trastuzumab
Measure: Median (Inter-Quartile Range); unit: SUVmax (g/mL)
Arm/Group | HER2+ Patients | HER2- Patients
Number analyzed (Participants) | 11 | 7
SUVmax (g/mL) | 7.0 [4.8 to 10.6] | 3.7 [3.0 to 4.7]
Statistical Analysis 1: Comparison: HER2+ Patients vs HER2- Patients; Test type: Other; p < 0.001, Wilcoxon rank-sum

2. Primary Outcome: Tumor Uptake of 64Cu-DOTA-trastuzumab After 48 Hours
Description: as for outcome 1
Time Frame: 48 hours after injection of 64 CU-DOTA-trastuzumab
Measure: Median (Inter-Quartile Range); unit: SUVmax (g/mL)
Arm/Group | HER2+ Patients | HER2- Patients
Number analyzed (Participants) | 11 | 7
SUVmax (g/mL) | 8.7 [5.7 to 13.0] | 4.6 [3.8 to 5.0]
Statistical Analysis 1: Comparison: HER2+ Patients vs HER2- Patients; Test type: Other; p < 0.001, Wilcoxon rank-sum

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 2 years and 9 months.
Arm/Group | HER2+ Patients | HER2- Patients
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/7
Other Adverse Events (participants affected / at risk) | 0/11 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT01093612/Prot_SAP_000.pdf